CLINICAL TRIAL: NCT05504928
Title: Effectiveness of a School-centered Primary and Secondary Prevention Program on Prevalence of Latent Rheumatic Heart Disease
Brief Title: Effectiveness of a School-centered Prevention Program on Prevalence of Latent Rheumatic Heart Disease
Acronym: NEPAL4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NEPAL4
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Rheumatic Heart Disease; Rheumatic Heart Disease in Children
Keywords: Rheumatic Heart Disease; Primary Prevention; Secondary Prevention; Screening
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Intervention Model Description: Interrupted time series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Implementation of a dedicated school nurse program (Experimental): School nurse program providing health care through assessment, intervention and follow-up of group A β-hemolytic streptococcal pharyngitis and facilitation of secondary antibiotic prophylaxis for children with latent rheumatic heart disease.
  Interventions: Other: School nurse program

INTERVENTIONS:
Other: School nurse program — School nurse program providing health care through assessment, intervention and follow-up of group A β-hemolytic streptococcal pharyngitis and facilitation of secondary antibiotic prophylaxis for children with latent rheumatic heart disease.

SUMMARY:
The overall objective is to evaluate the effectiveness of a school-centered primary and secondary prevention program on the prevalence of latent rheumatic heart disease among schoolchildren in Nepal, and to investigate the role of socioeconomic and environmental factors in the development and progression of rheumatic heart disease.

DETAILED DESCRIPTION:
Three in four children worldwide grow up in regions of the world where patterns of acute rheumatic fever and rheumatic heart disease are endemic and where rheumatic heart disease accounts for >300'000 deaths every year. Evidence from a systematic review and meta-analysis of 10 studies indicated an incidence of group A β-hemolytic streptococcal (GAHBS) pharyngitis among children in low- to upper-middle income countries of 10.8 per 100 child-years with considerable heterogeneity between individual reports.

Timely detection of GAHBS pharyngitis by use of rapid antigen detection tests and initiation of antibiotic treatment represents an effective target for primary prevention. Early stages of rheumatic heart disease manifest with morphologic or functional valvular changes that can only be detected with echocardiography and are therefore latent. Latent stages of rheumatic heart disease are reversible with timely initiation of secondary antibiotic prophylaxis. A school-centered approach provides an opportunity to provide equitable access to a primary and secondary prophylaxis program with the potential to substantially reduce the burden of rheumatic heart disease in endemic regions.

All children 5-16 years of age from Tulsi Secondary Boarding School in Tulsipur, Nepal, will be eligible for inclusion. Sociodemographic characteristics and will be collected by means of a standardized interview. In a study using an interrupted time series design, prevalence of latent rheumatic heart disease will be measured by means of transthoracic echocardiography before, and two and four years after implementation of a dedicated school nurse program providing health care through assessment, intervention and follow-up of GAHBS pharyngitis and facilitation of secondary antibiotic prophylaxis for children with latent rheumatic heart disease.

Investigators expect to find a decrease in prevalence of rheumatic heart disease after implementation of a dedicated school-centered prevention program primarily led by school nurses, and to identify sociodemographic and environmental factors associated with the development and progression of rheumatic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-16 years
* Attending Tulsi Secondary Boarding School in Tulsipur, Nepal.

Exclusion Criteria:

* Children / primary caregivers not providing informed consent to participate
* Children not attending Tulsi Secondary Boarding School in Tulsipur.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of definite or borderline Rheumatic Heart Disease | 4 years
  Prevalence of definite or borderline Rheumatic Heart Disease according to the criteria of the World Heart Federation as assessed by systematic echocardiographic screening

SECONDARY OUTCOMES:
Group A β-hemolytic streptococcal pharyngitis | 4 years
  Number of patients with group A β-hemolytic streptococcal pharyngitis within study participation
Acute rheumatic fever | 4 years
  Number of patients with acute rheumatic fever within study participation
Rheumatic heart disease | 4 years
  Number of patients with rheumatic heart disease within study participation
Adverse reactions to penicillin injections | 4 years
  Number of patients with adverse reactions to penicillin injections within study participation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Prof. Dr., Principal Investigator — Bern University Hospital
Locations (1):
- Tulsi Secondary Boarding School, Tulsi̇̄pur, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Marijon E, Mirabel M, Celermajer DS, Jouven X. Rheumatic heart disease. Lancet. 2012 Mar 10;379(9819):953-964. doi: 10.1016/S0140-6736(11)61171-9. PMID 22405798
- [Background] Watkins DA, Johnson CO, Colquhoun SM, Karthikeyan G, Beaton A, Bukhman G, Forouzanfar MH, Longenecker CT, Mayosi BM, Mensah GA, Nascimento BR, Ribeiro ALP, Sable CA, Steer AC, Naghavi M, Mokdad AH, Murray CJL, Vos T, Carapetis JR, Roth GA. Global, Regional, and National Burden of Rheumatic Heart Disease, 1990-2015. N Engl J Med. 2017 Aug 24;377(8):713-722. doi: 10.1056/NEJMoa1603693. PMID 28834488
- [Background] Pearce S, Bowen AC, Engel ME, de la Lande M, Barth DD. The incidence of sore throat and group A streptococcal pharyngitis in children at high risk of developing acute rheumatic fever: A systematic review and meta-analysis. PLoS One. 2020 Nov 18;15(11):e0242107. doi: 10.1371/journal.pone.0242107. eCollection 2020. PMID 33206687